CLINICAL TRIAL: NCT02720081
Title: A Phase-II, Randomized, Placebo-Controlled, Parallel-Group Clinical Trial to Study the Efficacy and Safety of MK-1029 in Adult Subjects With Persistent Asthma That is Uncontrolled While Receiving Montelukast.
Brief Title: Study of MK-1029 in Participants With Persistent Asthma That Cannot Be Controlled With Montelukast (MK-1029-015)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1029-015; 2015-005054-36 (EudraCT Number); MK-1029-015 (Other: Merck Registration Number); 163313 (Registry Identifier: JAPIC-CTI)
Record Dates: First submitted 2016-03-22; First posted 2016-03-25 (Estimated); Results first posted 2018-08-28 (Actual); Last update posted 2018-09-27 (Actual); Status verified 2018-08

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma | interventions — montelukast; Albuterol

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- MK-1029 150 mg + Montelukast 10 mg (Experimental): Participants receive single-blind MK-1029 Matching-image Placebo + open-label Montelukast 10 mg for a 2 to 4 week run-in period while discontinuing or tapering off asthma controller medications. Participants receive double-blind MK-1029 150 mg + Montelukast 10 mg for 6 weeks in the treatment period. Participants can use rescue medication during both periods as needed.
  Interventions: Drug: MK-1029 150 mg; Drug: Montelukast 10 mg; Drug: Albuterol/Salbutamol 90 mcg - 100 mcg per inhalation
- MK-1029 Placebo + Montelukast 10 mg (Placebo Comparator): Participants receive single-blind MK-1029 Matching-image Placebo + open-label Montelukast 10 mg for a 2 to 4 week run-in period while discontinuing or tapering off asthma controller medications. Participants receive double-blind MK-1029 Matching-image Placebo + Montelukast 10 mg for 6 weeks in the treatment period. Participants can use rescue medication during both periods as needed.
  Interventions: Drug: MK-1029 Matching-image Placebo; Drug: Montelukast 10 mg; Drug: Albuterol/Salbutamol 90 mcg - 100 mcg per inhalation

INTERVENTIONS:
Drug: MK-1029 150 mg — 150 mg tablet administered orally, once a day (QD), at bedtime
  Arms: MK-1029 150 mg + Montelukast 10 mg
Drug: MK-1029 Matching-image Placebo — Matching-image placebo tablet administered orally, QD, at bedtime
  Arms: MK-1029 Placebo + Montelukast 10 mg
Drug: Montelukast 10 mg — 10 mg tablet administered orally, QD, at bedtime
  Other Names: SINGULAIR®; Montelukast sodium
Drug: Albuterol/Salbutamol 90 mcg - 100 mcg per inhalation — 1 or 2 inhalations 4 times a day (QID) as needed (PRN) as a Rescue Medication

SUMMARY:
The purpose of this trial is to compare the safety, tolerability, and efficacy of adding MK-1029 to montelukast in adults with persistent asthma that is uncontrolled while receiving montelukast alone. Participants will have a specific genetic marker for clinical efficacy of MK-1029. The primary hypothesis is that when added to montelukast, treatment with MK-1029 is superior to placebo, as demonstrated by an increase in forced expiratory volume in one second (FEV1), measured as the average change from baseline at the end of Week 4 and Week 6 of treatment.

ELIGIBILITY:
Inclusion Criteria:

* Symptoms of persistent asthma for at least one year
* History of asthma treatments including "as-needed" inhaled short-acting beta-agonists (albuterol/salbutamol); stable doses of inhaled corticosteroids (ICS), combination ICS/long-acting (inhaled) Beta2-adrenergic agonist (LABA) and/or oral asthma controller(s)
* Must be able to discontinue or taper asthma controlling medications while receiving Montelukast
* No history of smoking or no smoking for at least 1 year, with a smoking history of no more than 10 pack-years
* Body Mass Index (BMI) of 15 kg/m^2 to 40 kg/m^2.
* Females must not be pregnant (negative serum human chorionic gonadotropin test) or breastfeeding and must not plan to become pregnant for the duration of the study, including the post-treatment follow-up period
* Women and male participants of reproductive potential must agree to use adequate contraception for the duration of the study

Exclusion Criteria:

* Evidence of another active pulmonary disorder such as bronchiectasis or chronic obstructive pulmonary disease (COPD)
* Unable to perform acceptable, repeatable spirometry
* History of myocardial infarction, congestive heart failure, or uncontrolled cardiac arrhythmia within 3 months of screening visit
* Major surgical procedure(s) within 4 weeks of screening visit
* Blood donation within 2 weeks of screening visit
* Treatment in an emergency room for asthma (within 4 weeks) or hospitalization for asthma or respiratory condition within 2 months of screening visit
* Evidence of active sinus disease within 2 weeks of screening visit
* Upper respiratory infection (viral or bacterial) within 1 month of screening visit
* History of a psychiatric disorder within 3 months of screening visit
* History of human immunodeficiency virus (HIV)
* Unstable disease of the ophthalmologic, neurological, hepatic, renal, connective tissue, genitourinary, gastrointestinal, cardiovascular or hematologic systems
* History of cancer (except for successfully treated basal and squamous cell carcinomas of the skin) within 5 years of screening visit
* Uncontrolled hypertension
* Participation in a clinical trial involving an investigational drug within 4 weeks of screening visit
* Hypersensitivity or intolerance to inhaled beta-agonists and/or leukotriene inhibitors or any of their ingredients, including lactose and galactose
* Known sensitivity to or has not had previous exposure to aspirin or non-steroidal anti-inflammatory drugs

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 142 (Actual)
Dates: Start 2016-05-11 (Actual); Primary Completion 2017-08-16 (Actual); Study Completion 2017-09-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: Yes
https://www.merck.com/clinical-trials/pdf/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | MK-1029 150 mg + Montelukast 10 mg | MK-1029 Placebo + Montelukast 10 mg
Started | 72 | 70
Treated | 70 | 69
Completed | 68 | 66
Not Completed | 4 | 4
Not completed — Adverse Event | 0 | 3
Not completed — Protocol Violation | 4 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | MK-1029 150 mg + Montelukast 10 mg | MK-1029 Placebo + Montelukast 10 mg | Total
Number analyzed (Participants) | 72 | 70 | 142
Age, Continuous [Mean (Standard Deviation); unit: Years] | 44.4 (12.1) | 42.2 (13.0) | 43.3 (12.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 41 | 46 | 87
  Male | 31 | 24 | 55
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 2 | 4
  Asian | 48 | 42 | 90
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 10 | 16 | 26
  More than one race | 12 | 10 | 22
  Unknown or Not Reported | 0 | 0 | 0
Pre beta-agonist (β-agonist) forced expiratory volume in one second (FEV1) Predicted [Mean (Standard Deviation); unit: Liter (L)] — If Week 0 measurement was not available, the last non-missing value before treatment was used as Baseline. Population: Analysis population consists of participants with pre β-agonist FEV1 predicted baseline data.
  Liter (L)
    number analyzed (Participants) | 70 | 69 | 139
    (all) | 2.251 (0.572) | 2.243 (0.631) | 2.247 (0.600)
C Alleles at the pre-specified single nucleotide polymorphism (SNP) [Count of Participants; unit: Participants] — Copies of C Alleles at the pre-specified SNP is the proposed genetic marker for response to MK-1029 for the treatment of asthma.
  Participants
    1 copy | 48 | 47 | 95
    2 copies | 24 | 23 | 47
Prior inhaled corticosteroid use [Count of Participants; unit: Participants]
  Yes | 52 | 54 | 106
  No | 20 | 16 | 36

OUTCOME MEASURES:

1. Primary Outcome: Baseline Pre-dose Forced Expiratory Volume in One Second (FEV1)
Description: FEV1 is the amount of air, measured in liters, forcibly exhaled in 1 second.
Time Frame: Before the first dose of study investigational product (Baseline)
Population: Analysis population consists of randomized participants who received at least 1 dose of study drug.
Measure: Mean (Standard Deviation); unit: Liter
Arm/Group | MK-1029 150 mg + Montelukast 10 mg | MK-1029 Placebo + Montelukast 10 mg
Number analyzed (Participants) | 70 | 69
Liter | 2.264 (0.566) | 2.234 (0.612)

2. Secondary Outcome: Percentage of Days With Worsening Asthma Average Over Weeks 3 to 6
Description: A day with worsening asthma was defined as any day during which any of the following occurred: a decrease from baseline in morning (AM) peak expiratory flow (PEF) of more than 20%; AM PEF less than 180 liters/minute (L/min); an increase in β-agonist use of more than 70% (and a minimum increase of at least 2 puffs); an increase from baseline in daytime asthma symptom score of more than 50%; overnight asthma symptom of: Awake "all night"; an asthma attack, as defined by any day when one or more of the following events due to asthma has occurred: corticosteroid use (systemic); unscheduled visit to the doctor or urgent care clinic; unscheduled visit to the emergency department; and/or hospitalization. Participants needed at least 80% of days with a complete diary during Weeks 3 to 6. A diary is considered complete if none of the above 6 components used to determine asthma worsening are missing.
Time Frame: Up to 4 weeks
Population: Analysis population consists of randomized participants who received at least 1 dose of study drug and had at least 80% of days with a complete diary during Weeks 3 to 6 (a diary is considered complete if none of the 6 components used to determine asthma worsening are missing).
Measure: Least Squares Mean (95% Confidence Interval); unit: Percentage of days
Arm/Group | MK-1029 150 mg + Montelukast 10 mg | MK-1029 Placebo + Montelukast 10 mg
Number analyzed (Participants) | 52 | 44
Percentage of days | 16.970 [10.115 to 23.826] | 21.746 [14.291 to 29.201]
Statistical Analysis 1: Comparison: MK-1029 150 mg + Montelukast 10 mg vs MK-1029 Placebo + Montelukast 10 mg; Test type: Superiority; p = 0.352, ANOVA; Terms for treatment, number of C alleles at the pre-specified SNP, and prior inhaled corticosteroid use; Difference in least squares means = -4.775, 95% CI 2-sided [-14.92 to 5.370]

3. Secondary Outcome: Percentage of Participants Who Experienced an Adverse Event (AE)
Description: An adverse event is defined as any untoward medical occurrence in a patient or clinical investigation participant administered a pharmaceutical product and which does not necessarily have to have a causal relationship with this treatment.
Time Frame: Up to 8 weeks
Population: Analysis population included all randomized participants who received at least 1 dose of study drug.
Measure: Number; unit: Percentage of participants
Arm/Group | MK-1029 150 mg + Montelukast 10 mg | MK-1029 Placebo + Montelukast 10 mg
Number analyzed (Participants) | 70 | 69
Percentage of participants | 25.7 | 26.1
Statistical Analysis 1: Comparison: MK-1029 150 mg + Montelukast 10 mg vs MK-1029 Placebo + Montelukast 10 mg; Test type: Other; Difference in percentages = -0.4, 95% CI 2-sided [-15.0 to 14.3] — Based on Miettinen & Nurminen

4. Secondary Outcome: Percentage of Participants Who Discontinued Study Drug Due to an AE
Description: as for outcome 3
Time Frame: Up to 6 weeks
Population: Analysis population included all randomized participants who received at least 1 dose of study drug.
Measure: Number; unit: Percentage of participants
Arm/Group | MK-1029 150 mg + Montelukast 10 mg | MK-1029 Placebo + Montelukast 10 mg
Number analyzed (Participants) | 70 | 69
Percentage of participants | 0.0 | 4.3
Statistical Analysis 1: Comparison: MK-1029 150 mg + Montelukast 10 mg vs MK-1029 Placebo + Montelukast 10 mg; Test type: Other; Difference in percentages = -4.3, 95% CI 2-sided [-12.1 to 1.0] — Based on Miettinen & Nurminen

5. Secondary Outcome: Change From Baseline in Alkaline Phosphatase (ALP) at Week 6
Description: Baseline was defined at Week 0. If Week 0 measurement is not available, the last non-missing value before treatment was used as Baseline.
Time Frame: Baseline and Week 6
Population: Analysis population includes all participants who received at least 1 dose of study drug and had non-missing change from baseline value at Week 6 for the analysis endpoint, ALP.
Measure: Mean (Standard Deviation); unit: IU/L
Arm/Group | MK-1029 150 mg + Montelukast 10 mg | MK-1029 Placebo + Montelukast 10 mg
Number analyzed (Participants) | 70 | 68
IU/L
  Baseline | 61.16 (19.05) | 67.96 (21.17)
  Change at Week 6 | -0.83 (7.68) | 0.44 (9.98)

6. Secondary Outcome: Change From Baseline in Alanine Aminotransferase (ALT) at Week 6
Description: as for outcome 5
Time Frame: Baseline and Week 6
Population: Analysis population includes all participants who received at least 1 dose of study drug and had non-missing change from baseline value at Week 6 for the analysis endpoint, ALT.
Measure: Mean (Standard Deviation); unit: IU/L
Arm/Group | MK-1029 150 mg + Montelukast 10 mg | MK-1029 Placebo + Montelukast 10 mg
Number analyzed (Participants) | 70 | 68
IU/L
  Baseline | 22.33 (12.75) | 19.35 (9.77)
  Change at Week 6 | -0.99 (9.84) | 0.34 (6.31)

7. Secondary Outcome: Change From Baseline in Aspartate Aminotransferase (AST) at Week 6
Description: as for outcome 5
Time Frame: Baseline and Week 6
Population: Analysis population includes all participants who received at least 1 dose of study drug and had non-missing change from baseline value at Week 6 for the analysis endpoint, AST.
Measure: Mean (Standard Deviation); unit: IU/L
Arm/Group | MK-1029 150 mg + Montelukast 10 mg | MK-1029 Placebo + Montelukast 10 mg
Number analyzed (Participants) | 70 | 67
IU/L
  Baseline | 23.53 (10.28) | 20.64 (7.62)
  Change at Week 6 | -0.09 (12.52) | 0.76 (7.67)

8. Secondary Outcome: Change From Baseline in Bilirubin at Week 6
Description: as for outcome 5
Time Frame: Baseline and Week 6
Population: Analysis population includes all participants who received at least 1 dose of study drug and had non-missing change from baseline value at Week 6 for the analysis endpoint, bilirubin.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | MK-1029 150 mg + Montelukast 10 mg | MK-1029 Placebo + Montelukast 10 mg
Number analyzed (Participants) | 70 | 68
mg/dL
  Baseline | 0.62 (0.25) | 0.54 (0.21)
  Change at Week 6 | -0.00 (0.25) | -0.01 (0.20)

9. Secondary Outcome: Change From Baseline in Eosinophil (Percent [%]) at Week 6
Description: as for outcome 5
Time Frame: Baseline and Week 6
Population: Analysis population includes all participants who received at least 1 dose of study drug and had non-missing change from baseline value at Week 6 for the analysis endpoint, eosinophil (%).
Measure: Mean (Standard Deviation); unit: Percent of White Blood Cells
Arm/Group | MK-1029 150 mg + Montelukast 10 mg | MK-1029 Placebo + Montelukast 10 mg
Number analyzed (Participants) | 69 | 68
Percent of White Blood Cells
  Baseline | 4.40 (4.54) | 3.58 (2.65)
  Change at Week 6 | 0.11 (4.29) | 0.51 (1.96)

10. Secondary Outcome: Change From Baseline in Neutrophil (%) at Week 6
Description: as for outcome 5
Time Frame: Baseline and Week 6
Population: Analysis population includes all participants who received at least 1 dose of study drug and had non-missing change from baseline value at Week 6 for the analysis endpoint, neutrophil (%).
Measure: Mean (Standard Deviation); unit: Percent of White Blood Cells
Arm/Group | MK-1029 150 mg + Montelukast 10 mg | MK-1029 Placebo + Montelukast 10 mg
Number analyzed (Participants) | 69 | 68
Percent of White Blood Cells
  Baseline | 59.13 (10.30) | 57.86 (10.48)
  Change at Week 6 | -1.32 (10.53) | 0.12 (9.11)

11. Secondary Outcome: Change From Baseline in Platelet Count at Week 6
Description: as for outcome 5
Time Frame: Baseline and Week 6
Population: Analysis population includes all participants who received at least 1 dose of study drug and had non-missing change from baseline value at Week 6 for the analysis endpoint, platelet count.
Measure: Mean (Standard Deviation); unit: 10^9 cells/L
Arm/Group | MK-1029 150 mg + Montelukast 10 mg | MK-1029 Placebo + Montelukast 10 mg
Number analyzed (Participants) | 68 | 68
10^9 cells/L
  Baseline | 256.85 (60.83) | 258.44 (70.23)
  Change at Week 6 | -4.97 (30.93) | 2.65 (29.44)

12. Secondary Outcome: Change From Baseline in White Blood Cell Count at Week 6
Description: as for outcome 5
Time Frame: Baseline and Week 6
Population: Analysis population includes all participants who received at least 1 dose of study drug and had non-missing change from baseline value at Week 6 for the analysis endpoint, white blood cell count.
Measure: Mean (Standard Deviation); unit: 10^9 cells/L
Arm/Group | MK-1029 150 mg + Montelukast 10 mg | MK-1029 Placebo + Montelukast 10 mg
Number analyzed (Participants) | 69 | 68
10^9 cells/L
  Baseline | 6.76 (2.55) | 6.53 (1.88)
  Change at Week 6 | -0.08 (2.00) | 0.09 (1.51)

13. Secondary Outcome: Change From Baseline in Hematocrit (%) at Week 6
Description: as for outcome 5
Time Frame: Baseline and Week 6
Population: Analysis population includes all participants who received at least 1 dose of study drug and had non-missing change from baseline value at Week 6 for the analysis endpoint, hematocrit (%).
Measure: Mean (Standard Deviation); unit: Percent
Arm/Group | MK-1029 150 mg + Montelukast 10 mg | MK-1029 Placebo + Montelukast 10 mg
Number analyzed (Participants) | 69 | 68
Percent
  Baseline | 42.79 (3.98) | 42.64 (4.62)
  Change at Week 6 | -0.10 (2.05) | -0.33 (1.86)

14. Secondary Outcome: Change From Baseline in Systolic Blood Pressure at Week 2
Description: Baseline was defined at Week 0. If Week 0 measurement was not available, the last non-missing value before treatment was used as Baseline.
Time Frame: Baseline and Week 2
Population: Analysis population includes all participants who received at least 1 dose of study drug and had non-missing change from baseline value at Week 2 for the analysis endpoint, systolic blood pressure.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | MK-1029 150 mg + Montelukast 10 mg | MK-1029 Placebo + Montelukast 10 mg
Number analyzed (Participants) | 70 | 69
mmHg
  Baseline | 118.89 (16.28) | 118.83 (15.64)
  Change at Week 2 | -1.61 (9.00) | -1.23 (10.79)

15. Secondary Outcome: Change From Baseline in Systolic Blood Pressure at Week 4
Description: as for outcome 14
Time Frame: Baseline and Week 4
Population: Analysis population includes all participants who received at least 1 dose of study drug and had non-missing change from baseline value at Week 4 for the analysis endpoint, systolic blood pressure.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | MK-1029 150 mg + Montelukast 10 mg | MK-1029 Placebo + Montelukast 10 mg
Number analyzed (Participants) | 68 | 67
mmHg
  Baseline | 119.40 (16.22) | 118.82 (15.88)
  Change at Week 4 | -2.13 (10.14) | -1.99 (11.45)

16. Secondary Outcome: Change From Baseline in Systolic Blood Pressure at Week 6
Description: as for outcome 14
Time Frame: Baseline and Week 6
Population: Analysis population includes all participants who received at least 1 dose of study drug and had non-missing change from baseline value at Week 6 for the analysis endpoint, systolic blood pressure.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | MK-1029 150 mg + Montelukast 10 mg | MK-1029 Placebo + Montelukast 10 mg
Number analyzed (Participants) | 68 | 66
mmHg
  Baseline | 119.40 (16.22) | 118.77 (16.00)
  Change at Week 6 | -0.34 (9.36) | -2.26 (11.11)

17. Secondary Outcome: Change From Baseline in Diastolic Blood Pressure at Week 2
Description: as for outcome 14
Time Frame: Baseline and Week 2
Population: Analysis population includes all participants who received at least 1 dose of study drug and had non-missing change from baseline value at Week 2 for the analysis endpoint, diastolic blood pressure.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | MK-1029 150 mg + Montelukast 10 mg | MK-1029 Placebo + Montelukast 10 mg
Number analyzed (Participants) | 70 | 69
mmHg
  Baseline | 74.40 (10.79) | 74.45 (10.49)
  Change at Week 2 | -1.31 (7.67) | -0.97 (6.88)

18. Secondary Outcome: Change From Baseline in Diastolic Blood Pressure at Week 4
Description: as for outcome 14
Time Frame: Baseline and Week 4
Population: Analysis population includes all participants who received at least 1 dose of study drug and had non-missing change from baseline value at Week 4 for the analysis endpoint, diastolic blood pressure.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | MK-1029 150 mg + Montelukast 10 mg | MK-1029 Placebo + Montelukast 10 mg
Number analyzed (Participants) | 68 | 67
mmHg
  Baseline | 74.60 (10.88) | 74.42 (10.49)
  Change at Week 4 | -1.56 (7.71) | -1.60 (8.01)

19. Secondary Outcome: Change From Baseline in Diastolic Blood Pressure at Week 6
Description: as for outcome 14
Time Frame: Baseline and Week 6
Population: Analysis population includes all participants who received at least 1 dose of study drug and had non-missing change from baseline value at Week 6 for the analysis endpoint, diastolic blood pressure.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | MK-1029 150 mg + Montelukast 10 mg | MK-1029 Placebo + Montelukast 10 mg
Number analyzed (Participants) | 68 | 66
mmHg
  Baseline | 74.60 (10.88) | 74.29 (10.51)
  Change at Week 6 | -1.18 (8.30) | -0.95 (7.71)

20. Secondary Outcome: Change From Baseline in Heart Rate at Week 2
Description: as for outcome 14
Time Frame: Baseline and Week 2
Population: Analysis population includes all participants who received at least 1 dose of study drug and had non-missing change from baseline value at Week 2 for the analysis endpoint, heart rate.
Measure: Mean (Standard Deviation); unit: beats/min
Arm/Group | MK-1029 150 mg + Montelukast 10 mg | MK-1029 Placebo + Montelukast 10 mg
Number analyzed (Participants) | 70 | 69
beats/min
  Baseline | 73.21 (10.96) | 74.20 (10.03)
  Change at Week 2 | -0.60 (7.84) | 0.45 (9.38)

21. Secondary Outcome: Change From Baseline in Heart Rate at Week 4
Description: as for outcome 14
Time Frame: Baseline and Week 4
Population: Analysis population includes all participants who received at least 1 dose of study drug and had non-missing change from baseline value at Week 4 for the analysis endpoint, heart rate.
Measure: Mean (Standard Deviation); unit: beats/min
Arm/Group | MK-1029 150 mg + Montelukast 10 mg | MK-1029 Placebo + Montelukast 10 mg
Number analyzed (Participants) | 68 | 67
beats/min
  Baseline | 73.25 (11.12) | 73.96 (10.01)
  Change at Week 4 | -1.82 (9.18) | 1.40 (9.38)

22. Secondary Outcome: Change From Baseline in Heart Rate at Week 6
Description: as for outcome 14
Time Frame: Baseline and Week 6
Population: Analysis population includes all participants who received at least 1 dose of study drug and had non-missing change from baseline value at Week 6 for the analysis endpoint, heart rate.
Measure: Mean (Standard Deviation); unit: beats/min
Arm/Group | MK-1029 150 mg + Montelukast 10 mg | MK-1029 Placebo + Montelukast 10 mg
Number analyzed (Participants) | 68 | 66
beats/min
  Baseline | 73.25 (11.12) | 73.80 (10.01)
  Change at Week 6 | -0.84 (8.82) | 1.06 (10.10)

23. Secondary Outcome: Change From Baseline in Respiratory Rate at Week 2
Description: as for outcome 14
Time Frame: Baseline and Week 2
Population: Analysis population includes all participants who received at least 1 dose of study drug and had non-missing change from baseline value at Week 2 for the analysis endpoint, respiratory rate.
Measure: Mean (Standard Deviation); unit: breaths/min
Arm/Group | MK-1029 150 mg + Montelukast 10 mg | MK-1029 Placebo + Montelukast 10 mg
Number analyzed (Participants) | 70 | 69
breaths/min
  Baseline | 16.40 (2.61) | 17.23 (3.78)
  Change at Week 2 | -0.30 (1.93) | -1.17 (3.64)

24. Secondary Outcome: Change From Baseline in Respiratory Rate at Week 4
Description: as for outcome 14
Time Frame: Baseline and Week 4
Population: Analysis population includes all participants who received at least 1 dose of study drug and had non-missing change from baseline value at Week 4 for the analysis endpoint, respiratory rate.
Measure: Mean (Standard Deviation); unit: breaths/min
Arm/Group | MK-1029 150 mg + Montelukast 10 mg | MK-1029 Placebo + Montelukast 10 mg
Number analyzed (Participants) | 68 | 67
breaths/min
  Baseline | 16.43 (2.60) | 17.18 (3.82)
  Change at Week 4 | -0.12 (2.58) | -0.97 (3.24)

25. Secondary Outcome: Change From Baseline in Respiratory Rate at Week 6
Description: as for outcome 14
Time Frame: Baseline and Week 6
Population: Analysis population includes all participants who received at least 1 dose of study drug and had non-missing change from baseline value at Week 6 for the analysis endpoint, respiratory rate.
Measure: Mean (Standard Deviation); unit: breaths/min
Arm/Group | MK-1029 150 mg + Montelukast 10 mg | MK-1029 Placebo + Montelukast 10 mg
Number analyzed (Participants) | 68 | 66
breaths/min
  Baseline | 16.43 (2.60) | 17.20 (3.84)
  Change at Week 6 | -0.09 (2.30) | -1.17 (3.20)

26. Primary Outcome: Average Change From Baseline in Pre-dose FEV1 at Week 4 and Week 6
Description: FEV1 is the amount of air, measured in liters, forcibly exhaled in 1 second. Pulmonary function tests were to be performed by participants in the morning before dosing. Data presented represents the average change from baseline at Week 4 and Week 6.
Time Frame: Before the first dose (Baseline) and at the end of Weeks 4 and 6 of treatment
Population: Analysis population consists of randomized participants who received at least 1 dose of study drug.
Measure: Least Squares Mean (95% Confidence Interval); unit: Liter
Arm/Group | MK-1029 150 mg + Montelukast 10 mg | MK-1029 Placebo + Montelukast 10 mg
Number analyzed (Participants) | 70 | 69
Liter | 0.152 [0.088 to 0.217] | 0.046 [-0.020 to 0.111]
Statistical Analysis 1: Comparison: MK-1029 150 mg + Montelukast 10 mg vs MK-1029 Placebo + Montelukast 10 mg; Test type: Superiority; p = 0.023, Constrained longitudinal data analysis; Terms for treatment, time, interaction of time by treatment, number of C alleles at the pre-specified SNP, and prior inhaled corticosteroid use; Difference in least squares means = 0.107, 95% CI 2-sided [0.015 to 0.199]

ADVERSE EVENTS:
Time Frame: Up to 8 weeks
Description: Analysis population included all randomized participants who received at least 1 dose of study drug.
Arm/Group | MK-1029 150 mg + Montelukast 10 mg | MK-1029 Placebo + Montelukast 10 mg
All-Cause Mortality (participants affected / at risk) | 0/70 | 0/69
Serious Adverse Events (participants affected / at risk) | 0/70 | 1/69
Other Adverse Events (participants affected / at risk) | 6/70 | 9/69
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MK-1029 150 mg + Montelukast 10 mg (N=70) | MK-1029 Placebo + Montelukast 10 mg (N=69)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MK-1029 150 mg + Montelukast 10 mg (N=70) | MK-1029 Placebo + Montelukast 10 mg (N=69)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 4 (5)
Viral upper respiratory tract infection (Infections and infestations) | 4 (4) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 8 (8)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor must have the opportunity to review all proposed abstracts, manuscripts or presentations regarding this trial 45 days prior to submission for publication/presentation. Any information identified by the Sponsor as confidential must be deleted prior to submission; this confidentiality does not include efficacy and safety results.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-03-03): https://cdn.clinicaltrials.gov/large-docs/81/NCT02720081/Prot_SAP_000.pdf